CLINICAL TRIAL: NCT00257426
Title: A Phase II Study of Octreotide Acetate for the Treatment of Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: Octreotide in Treating Patients With Locally Advanced or Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0221; UNC-LCCC-0221; CDR0000561597 (Other: PDQ number)
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Octreotide

INTERVENTIONS:
Drug: octreotide acetate — 200mcg,3 times per day, 7 days per week, up to 36 weeks
  Other Names: Sandostatin

SUMMARY:
RATIONALE: Octreotide may stop or slow the growth of tumor cells and may be an effective treatment for liver cancer.

PURPOSE: This phase II trial is studying how well octreotide works in treating patients with locally advanced or metastatic liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To verify that long-acting somatostatin analog octreotide (Sandostatin LAR) depot will extend median survival from 5 months to 8.75 months in patients with locally advanced or metastatic hepatocellular carcinoma with a CLIP score of 3 or more.

Secondary

* To document tolerability of this drug in this patient population.

OUTLINE: Patients are stratified according to underlying degree of liver disease as defined by CLIP score classification.

Patients receive short-acting octreotide subcutaneously three times daily on days 1-21 OR days 1-28. If the patient tolerates short-acting octreotide, the first dose of long-acting octreotide (Sandostatin LAR) depot will be given intramuscularly beginning on day 8 OR day 15. Treatment with long-acting octreotide repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After the completion of study treatment, patients are followed monthly for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed or recurrent hepatocellular carcinoma (HCC) as defined by tissue biopsy OR alpha fetoprotein (AFP) > 1,000 ng/mL with compatible mass on CT scan or MRI

  * Recurrence of previously resected HCC will not require tissue confirmation if there is clear radiographic recurrence, in the judgment of the investigator
* Locally advanced OR metastatic disease
* Unmeasurable disease allowed if initial diagnosis was made according to the above criteria and/or recurrence has been confirmed by tissue biopsy or radiological imaging
* CLIP score ≥ 3
* Not a candidate for surgical resection or liver transplant
* Not a candidate for loco-regional therapy (e.g., ablation, embolization, hepatic arterial infusion therapy), but could have received such therapy in the past
* No fibrolamellar HCC
* No clinically apparent central nervous system metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 8 weeks
* Karnofsky performance status 60-100%
* Hemoglobin ≥ 8.5 g/dL
* Platelet count ≥ 50,000/mm³
* Total bilirubin ≤ 5.0 mg/dL
* AST or ALT ≤ 5 times upper limit of normal (ULN)
* Creatinine ≤ 2 times ULN
* PT ≤ 28
* INR ≤ 2.5
* No active variceal bleeding within the past 3 months
* No encephalopathy grade 3-4
* No ongoing ethanol or intravenous drug abuse
* Not pregnant or breast feeding

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Any number of prior therapies (e.g., chemotherapy, resection, embolization, or radiofrequency/ethanol ablation therapy) allowed
* No concurrent chemotherapy, radiotherapy, or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-07; Primary Completion 2007-02 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Median survival | 6 months

SECONDARY OUTCOMES:
number of subjects with toxicities | 6 months
  Toxicities will be graded using the NCI's Common Toxicity Criteria, Version 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Bert H. O'Neil, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- The University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States